CLINICAL TRIAL: NCT00002581
Title: PROTOCOL FOR THE SCOTTISH POSTMENOPAUSAL CHEMO-ENDOCRINE TRIAL
Brief Title: Tamoxifen With or Without Combination Chemotherapy in Treating Postmenopausal Women With Operable Invasive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063696; SCTN-BR9402; EU-94003; UKCCCR-ABC/BR9402
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Fluorouracil; Methotrexate; Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fluorouracil
Drug: methotrexate
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Combining combination chemotherapy with hormone therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of tamoxifen with or without combination chemotherapy in treating postmenopausal women with stage I or stage II breast cancer that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the potential benefits of adjuvant tamoxifen with or without cyclophosphamide, methotrexate, and fluorouracil (CMF) in postmenopausal women with stage I-IIIA, unilateral, invasive breast cancer.

OUTLINE: This is a randomized study, multicenter study. Patients are stratified according to nodal status (positive vs negative or unknown) and hospital region. Patients undergo surgical resection with or without local radiotherapy, as appropriate. Radiotherapy begins within 8 weeks of surgery for patients randomized to arm I and within 4 weeks after completion of chemotherapy for patients randomized to arm II. Patients are randomized to 1 of 2 treatment arms, preferably within 2 weeks after surgery. Arm I: Beginning within 4 weeks after surgery, patients receive oral tamoxifen daily. Treatment continues for 5 years. Arm II: Beginning within 4 weeks after surgery, patients receive tamoxifen as in arm I and cyclophosphamide IV, methotrexate IV, and fluorouracil IV on day 1 (CMF). Chemotherapy continues every 3 weeks for 6 courses. Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unilateral, invasive breast cancer Stage T0-3, N0-1, M0 No evidence of distant disease, including ipsilateral supraclavicular node enlargement unless proven benign No carcinoma in situ alone, including Paget's disease of the nipple without underlying invasion No evidence of distant disease, including ipsilateral supraclavicular node enlargement unless proven benign No history of pure carcinoma in situ in either breast Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 70 and under Sex: Female Menopausal status: Postmenopausal, defined by 1 of the following criteria: Last menstrual period more than 1 year before initial surgery Any age with prior bilateral oophorectomy (for nonmalignant reason) Age 50 and over with prior hysterectomy (for nonmalignant reason) without oophorectomy If at variance with the above definitions, hormonal assays in postmenopausal range take precedence Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other serious illness No other prior invasive malignancy except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1993-06

CONTACTS AND LOCATIONS:
Overall Officials: W.D. George, MD, MS, FRCS, Study Chair — University of Glasgow
Locations (9):
- United Kingdom (9):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - University of Glasgow, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Ayr Hospital, Ayr
  - Falkirk Royal Infirmary, Falkirk